CLINICAL TRIAL: NCT05054517
Title: The Use of Oral Glutamine in Patients With Thoracic and Upper Aerodigestive Malignancies Who Undergo Radiotherapy: Results of a Prospective Observational Study
Brief Title: Oral Glutamine and Thoracic/Upper Aerodigestive Tumors Radiation Toxicity
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Nikolaos Drakoulis, MD, Prof. Dr., National and Kapodistrian University of Athens
Other Study IDs: Athens Medical 2281/26-04-2013
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Biopsy Confirmed Head and Neck Cancer and Tumors of the Chest
Keywords: Glutamine; chest tumors; lung cancer; head and neck cancer; clinical studies; human subjects
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms | interventions — Glutamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Glutamine — Oral Supplement

SUMMARY:
PROTOCOL FOR PREVENTIVE ADMINISTRATION OF GLUTAMINE TO AVOID RADIATE SIDE EFFECTS IN PATIENTS UNDER RADIOTHERAPY IN THE CHEST AND HEAD & NECK

PURPOSE OF THE STUDY

The purpose of the protocol is to study the acute and distant toxicity of the mucosa of the oral cavity and esophagus after radiotherapy for head-neck and tumors of the chest. Radiation therapy in all cases is a three-dimensional conformal technique with a linear accelerator.

INCLUSION CRITERIA

Patients undergoing radiotherapy with or without concomitant chemotherapy for Ca nasopharynx, hypopharynx, palate, tonsils, mouth base, parotid, tongue, cervix and esophagus as well as mediastinal and lung cancer.

EXCLUSION CRITERIA

Patients with psychiatric problems and inability to cooperate, as well as patients with gluten intolerance, as well as patients with hepatic encephalopathy or hyperammonemia, are excluded from the study.

METHODS

Oral glutamine administration starting 4 days before the start of radiotherapy and for a total of 3 months. The preparation is dissolved in water and taken orally 4 hours before radiotherapy and 4 hours before dinner.

FOLLOW UP

Immediately after completion of radiotherapy at 3, 6 and 12 months, orthoscopy (on symptoms) and oral mucosal examination will be performed on patients who have undergone cervical and mediastinal radiotherapy and their evaluation based on the EORTC-RTOG scale.

REFERENCES

1. Anderson PM, Schroeder G, Skubitz KM. "Oral glutamine reduces the duration and severity of stomatitis after cytotoxic cancer chemotherapy". Cancer: 1998; 83: 1433-1439.
2. Cerchietti LC, Navigante AH, Lutteral MA, Castro MA, Kirchuk R, Bonomi M et al. "Double-blinded, placebo-controlled trial on intravenous L-alanyl-L-glutamine in the incidence of oral mucosis following chemotherapy in patients with head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2006 Aug 1; 65 (5): 1330-7.
3. Peterson DE, Jones JB, Petit RG 2nd. "Randomized, placebo-controlled trial of Saforis for prevention and treatment of oral mucositis in breast cancer patients receiving anthracycline-based chemotherapy. Cancer. 2007 Jan 15; 109(2): 322-31.
4. Kozelsky TF, Meyers GE, Sloan JA, Shanahan TG, Dick SJ et al; North Central Cancer Treatment Group. Mayo Clinic "Phase III double-blind study of glutamine versus placebo for the prevention of acute diarrhea in patients receiving pelvic radiation therapy". J Clin Oncol 2003 May 1; 21 (9):1669-74.
5. Topkan E, Yavuz MN, et al "Prevention of acute radiation-induced esophagitis with glutamine in non-small cell lung cancer patients treated with radiotherapy: Evaluation of clinical and dosimetric parameters". Lung Cancer, 2008 August 6.
6. Ismael Membrive Conejo, Ana Reig Castillejo, Nuria Rodriguez de Dios, Palmira Foro Arnalot, Javier Sanz Latiesas, et al: "Prevention of acute radiation enteritis: efficacy and tolerance of glutamine". Clinical and Translational Oncology. Vol 13, Number 10 (2011), 760-763, DOI: 10.1007/st 2094-011-0729-3.
7. Yoshida S, Kaibara A, Ishibashi N, Shirouzu K. "Glutamine supplementation in cancer patients" Nutrition. 2001: 17:766-768.
8. Klimberg SV, McClellan Jl. "Glutamine, cancer and its therapy. Am J Surg. 1996;172: 172:418-424.
9. Rouse K, Nwokedi E, Woodliff JE, Epstein J, Klimberg VS. "Glutamine enhances selectivity of chemotherapy through changes in glutathione metabolism. Ann Surg. 1995; 221:420-426.
10. Baxevanis CN, Reclos GJ, Grittapis AD et al "Elevated PGE2 production by monocytes is responsible for the depressed levels of NK&LAK cell function in patients with breast cancer" Cancer. 1993; 12:491-501.
11. Erdem NZ, Yasti AC, Atli M, et al. "The effects of perioperative oral enteral support with glutamine added elemental formulas in patients with gastrointestinal cancers: a prospective randomized clinical study. Nutr Res.2002:22:977-988.
12. Berk L, James J, Schwartz A, Hug E, Mahadevan A, Samuels M et al. "A randomized, double-blind, placebo-controlled trial of a beta hydroxyl beta-methyl butyrate, glutamine, and arginine mixture for the treatment of cancer cachexia". Support Care Cancer. 2008 Oct; 16 (10): 1179-88. Epub 2008 Feb 22.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radiotherapy with or without concomitant chemotherapy for Ca nasopharynx, hypopharynx, palate, tonsils, mouth base, parotid, tongue, cervix and esophagus as well as mediastinal and lung cancer.

Exclusion Criteria:

* Patients with psychiatric problems and inability to cooperate, as well as patients with gluten intolerance, as well as patients with hepatic encephalopathy or hyperammonemia are excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 72 patients with biopsy-diagnosed T&UAM were prospectively recruited. The mean age of patients was 65.6 ± 1.2 years, ranging between 54 and 77 years. Most participants were male (n=54, 75%).
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoints were the incidence of grade 2 or greater in the observed toxicities, weight loss and the need for analgesic therapy | one month

SECONDARY OUTCOMES:
The secondary endpoint was the length of the irradiated esophagus from radiotherapy (RT) treatment planning correlated with the use of opioids as analgesics. | one month

IPD SHARING:
Plan to Share IPD: No
no availability of any data

REFERENCES:
- [Derived] Papanikolopoulou A, Syrigos N, Vini L, Papasavva M, Lazopoulos G, Kteniadakis S, Spandidos DA, Charpidou A, Drakoulis N. Use of oral glutamine in radiation-induced adverse effects in patients with thoracic and upper aerodigestive malignancies: Results of a prospective observational study. Oncol Lett. 2022 Jan;23(1):19. doi: 10.3892/ol.2021.13137. Epub 2021 Nov 16. PMID 34858523